CLINICAL TRIAL: NCT00469105
Title: Improving Care for Primary Care Patients With Diabetes and Poor Literacy and Numeracy Skills
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); American Diabetes Association (Other); Pfizer (Industry)
Responsible Party: Russell Rothman, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 7-04-NN-16 (ADA); Vanderbilt IRB: 040387; UNC IRB: 06-0535
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Diabetes Education; Health Literacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Control Arm receives standard diabetes disease management
  Interventions: Behavioral: Control Group
- Intervention Arm (Experimental): Receives numeracy/literacy sensitive diabetes management
  Interventions: Behavioral: Literacy/Numeracy oriented educational intervention

INTERVENTIONS:
Behavioral: Literacy/Numeracy oriented educational intervention — Receives comprehensive literacy/num sensitive diabetes care
  Arms: Intervention Arm
Behavioral: Control Group — Receives standard diabetes disease management
  Arms: Control

SUMMARY:
The aim of this research will be to perform a small randomized controlled trial (RCT) of a new diabetes educational intervention that teaches self-management skills that compensate for poor numeracy skills among a sample of primary care patients with type 2 diabetes and low literacy and/or numeracy.

DETAILED DESCRIPTION:
Results of the National Adult Literacy Survey (NALS) suggest that over 90 million adult Americans have poor quantitative skills. Numeracy, the ability to understand and use numbers and math skills in daily life, may be particularly important to patients with diabetes because caring for diabetes often requires self-management skills that rely on the daily application of math skills, such as counting carbohydrates, interpreting blood glucose monitoring, applying sliding scale insulin regimens, and calculating insulin to carbohydrate ratios. Presumably diabetes patients with poor numeracy have more difficulty with self-management and are at risk for poorer clinical outcomes, but to date, there are no published studies that rigorously examine the role of numeracy in diabetes. We have recently completed the initial development of a new scale to measure numeracy in patients with diabetes: the Diabetes Numeracy Test (DNT).

The aim of this research will be to perform a small randomized controlled trial (RCT) of a new diabetes educational intervention that teaches self-management skills that compensate for poor literacy and numeracy skills among a sample of patients with type 2 diabetes and low numeracy or literacy skills. We hypothesize that a group of patients with poor literacy and/or numeracy who are taught self-management skills that accommodate their poor numeracy will have: (1) improved treatment satisfaction and perceived self-efficacy, (2) improved performance in self-management tasks, and (3) improved glycemic control compared to a control group that receives usual education and care.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Type 2 Diabetes
2. most recent A1C >= 7.5%
3. Referred to the Diabetes Care Program for diabetes care
4. Age 18-85; 5. English Speaking.

Exclusion Criteria:

1. Patients with corrected visual Acuity >20/50 using a Rosenbaum Pocket Vision Screener
2. Patients with a diagnosis of significant dementia, psychosis, or blindness.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
A1C | 3 and 6 months

SECONDARY OUTCOMES:
Patient self-management behaviors | 3 and 6 months
Patient knowledge | 6 months
Patient satisfaction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robb Malone, PharmD, Principal Investigator — University of North Carolina, Chapel Hill; Russell L Rothman, MD MPP, Principal Investigator — Vanderbilt University
Locations (1):
- University of North Carolina at Chapel Hill, General Medicine Clinic, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Cavanaugh K, Wallston KA, Gebretsadik T, Shintani A, Huizinga MM, Davis D, Gregory RP, Malone R, Pignone M, DeWalt D, Elasy TA, Rothman RL. Addressing literacy and numeracy to improve diabetes care: two randomized controlled trials. Diabetes Care. 2009 Dec;32(12):2149-55. doi: 10.2337/dc09-0563. Epub 2009 Sep 9. PMID 19741187